CLINICAL TRIAL: NCT05601596
Title: ROSE II: Pilot Study to Analyze Menstrual Blood to Predict Endometriosis
Brief Title: Research OutSmarts Endometriosis II Study
Acronym: ROSE2
Status: Enrolling by invitation | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Peter Gregersen, Professor and Director, Robert S. Boas Center for Genomics and Human Genetics, Northwell Health
Other Study IDs: 22-0346
Record Dates: First submitted 2022-08-04; First posted 2022-11-01 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Endometriosis
Keywords: Diagnosis
MeSH Terms: conditions — Endometriosis; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Menstrual effluent sample Optional peripheral blood sample 1 x 10 ml EDTA tube
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Participant: Having No symptoms of Endo. Provide Menstrual samples.
  Interventions: Diagnostic Test: Analysis of menstrual blood to predict endometriosis
- Symptomatic participant: Having symptoms of Endo and heading to diagnostic surgery as part of their standard of care (referred).
  Interventions: Diagnostic Test: Analysis of menstrual blood to predict endometriosis

INTERVENTIONS:
Diagnostic Test: Analysis of menstrual blood to predict endometriosis — Menstrual blood from controls and symptomatic cases will be analyzed using single cell RNA-sequencing to develop a panel of biomarkers that can be developed into a screening test or diagnostic test for endometriosis.

SUMMARY:
This product will be used as a diagnostic test to screen for the likelihood of endometriosis in menstruating adults with symptoms suggestive of endometriosis. The purpose of the test will be to guide clinical decisions regarding: 1) whether to undergo diagnostic laparoscopy to confirm the presence of endometriosis (currently, the gold standard for diagnosing endometriosis) and/or 2) how to guide the choice of hormonal or other therapies to treat symptoms of endometriosis.

DETAILED DESCRIPTION:
Endometriosis is a chronic, complex, and common gynecologic disorder characterized by the growth of endometrial-like tissues outside of the uterus that is accompanied by inflammation. One of the most frustrating problems for those with endometriosis is the long delay before being diagnosed, which can be up to 7-10 years. One of the reasons for this delay is that definitive diagnosis requires invasive surgery (Tomassetti et al, 2021 PMID: 34690084). There are no approved non-invasive methods for predicting endometriosis. This study will assess the analysis of fresh menstrual blood as a non-invasive predictor of endometriosis. This approach is based on the numerous reports documenting the differences in the endometrium of women with and without endometriosis; this endometrium is shed each month as menstrual blood which can be easily collected and analyzed. Through this prospective, non-interventional pilot study the investigators propose to collect and analyze menstrual blood from healthy controls without chronic symptoms of endometriosis and symptomatic women who have significant and chronic symptoms suggestive of endometriosis and are considered by their healthcare providers to be candidates for diagnostic laparoscopic surgery in the coming months (as part of their standard care). Menstrual blood from controls and symptomatic cases will be analyzed using single cell RNA-sequencing to develop a panel of biomarkers that can be developed into a screening test or diagnostic test for endometriosis.

The primary objectives of this study are to confirm the results of our recent single cell RNA sequencing (scRNA-Seq) analysis of menstrual effluent obtained from healthy controls vs. endometriosis (and symptomatic subjects) obtained through IRB 13-376 and to develop a screening/ diagnostic algorithm (menstrual global (MG) score) based on the data to be used to predict endometriosis in symptomatic patients.

The secondary objective is to assess the reproducibility of the scRNA-Sequencing data using menstrual blood collected across different menstrual cycles among a subset of controls and/or cases (symptomatic patients).

There are no existing commercially available products for the diagnostic analysis of cells or tissues present in menstrual effluent for endometriosis or any other condition. To our knowledge this is no commercially available product for predicting endometriosis using peripheral blood or other biological specimens (other than the analysis of ectopic endometriosis lesions themselves). Currently, definitive diagnosis of endometriosis requires laparoscopic surgery and pathological analysis of the removed ectopic lesions.

ELIGIBILITY:
Inclusion Criteria:

For All

* 18 to 40 year old menstruating women (continue to get cycles)
* More than a light menstrual flow (light flow is soaking less than 1 thin pad or light tampon in 4 hours at peak flow)
* Willingness to provide two menstrual samples across two separate menstrual cycles.
* Willingness to provide a DNA sample (obtained via menstrual blood or cheek swab)

For Controls:

•General Absence of *symptoms suggestive of endometriosis which includes: 1-Chronic pelvic pain 2-Painful menses 3-Pain during intercourse 4-Pain going to the bathroom 5-Abdominal bloating (BUT MUST NOT Include): 6-Report of missed days of work, school, athletic,social and/or other activities due to related pain and discomfort

For Symptomatic:

* Consistently Experiencing chronic symptoms of endometriosis*
* Without definitive diagnosis
* Seeking physician evaluation (considered by physician to be a candidate for laproscopic surgery
* Willingness to provide one of the menstrual samples PRIOR to planned surgery
* Surgical and pathological confirmation of endo (or NOT)

Exclusion Criteria:

For All:

* under age 18 or over 40 years
* Unable/unwilling to provide a menstrual sample
* Light menstrual flow (light flow is soaking less than 1 thin pad or light tampon in 4 hours at peak flow)
* Diagnosed with endometriosis

CONTROL:

* More than 1 symptom of endometriosis*
* Report of missed days of work, school, athletic, social and/or other activities due to related pain and discomfort

Symptomatic:

Unable to provide a menstrual sample prior to surgery

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The cohort will enroll a total of 185 menstruating individuals in total; 80 control subjects who self-report the general absence of symptoms of endometriosis and 105 symptomatic cases who report chronic symptoms* of endometriosis but who have not yet been diagnosed and are seeking physician evaluation for their symptoms.
Sampling Method: Probability Sample
Enrollment: 185 (Estimated)
Dates: Start 2022-05-27 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
ROSE II: Pilot study to analyze menstrual blood to predict endometriosis | 2 years
  The investigators will utilize single cell RNA sequencing analysis of stromal cells and uNK cells in menstrual effluent in order to define cellular and gene expression phenotypes that have been shown to be highly correlated with the presence of endometriosis

SECONDARY OUTCOMES:
ROSE II: Pilot study to assess the progesterone sensitivity or resistance of cultured endometrial stromal cells | 2 years
  The investigators will assess the response of endometrial stromal cells in menstrual blood to in vitro progesterone exposure using measurements of insulin growth factor binding protein 1 (IGFBP1) and prolactin (PRL).

CONTACTS AND LOCATIONS:
Overall Officials: Peter K Gregersen, MD, Principal Investigator — Northwell Health; Christine N Metz, PhD, Principal Investigator — Northwell Health
Locations (1):
- Feinstein Institutes/Northwell health, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
The PIs on the study will determine with whom the de-identified samples will be shared. If we share any samples with other researchers, then we will remove all identifiers such as name or date of birth before sharing them.

REFERENCES:
- [Background] Aghajanova L, Giudice LC. Molecular evidence for differences in endometrium in severe versus mild endometriosis. Reprod Sci. 2011 Mar;18(3):229-51. doi: 10.1177/1933719110386241. Epub 2010 Nov 9. PMID 21063030
- [Background] Ballard K, Lowton K, Wright J. What's the delay? A qualitative study of women's experiences of reaching a diagnosis of endometriosis. Fertil Steril. 2006 Nov;86(5):1296-301. doi: 10.1016/j.fertnstert.2006.04.054. PMID 17070183
- [Background] Brosens I, Brosens JJ, Benagiano G. The eutopic endometrium in endometriosis: are the changes of clinical significance? Reprod Biomed Online. 2012 May;24(5):496-502. doi: 10.1016/j.rbmo.2012.01.022. Epub 2012 Jan 31. PMID 22417665
- [Background] Bulun SE, Cheng YH, Yin P, Imir G, Utsunomiya H, Attar E, Innes J, Julie Kim J. Progesterone resistance in endometriosis: link to failure to metabolize estradiol. Mol Cell Endocrinol. 2006 Mar 27;248(1-2):94-103. doi: 10.1016/j.mce.2005.11.041. Epub 2006 Jan 10. PMID 16406281
- [Background] Chehna-Patel N, Sachdeva G, Gajbhiye R, Warty N, Khole V. "Spot"-ting differences between the ectopic and eutopic endometrium of endometriosis patients. Fertil Steril. 2010 Nov;94(6):1964-71, 1971.e1. doi: 10.1016/j.fertnstert.2010.01.048. Epub 2010 Mar 16. PMID 20236630
- [Background] Drury JA, Parkin KL, Coyne L, Giuliani E, Fazleabas AT, Hapangama DK. The dynamic changes in the number of uterine natural killer cells are specific to the eutopic but not to the ectopic endometrium in women and in a baboon model of endometriosis. Reprod Biol Endocrinol. 2018 Jul 18;16(1):67. doi: 10.1186/s12958-018-0385-3. PMID 30021652
- [Background] Dunselman GA, Vermeulen N, Becker C, Calhaz-Jorge C, D'Hooghe T, De Bie B, Heikinheimo O, Horne AW, Kiesel L, Nap A, Prentice A, Saridogan E, Soriano D, Nelen W; European Society of Human Reproduction and Embryology. ESHRE guideline: management of women with endometriosis. Hum Reprod. 2014 Mar;29(3):400-12. doi: 10.1093/humrep/det457. Epub 2014 Jan 15. PMID 24435778
- [Background] Johnston JL, Reid H, Hunter D. Diagnosing endometriosis in primary care: clinical update. Br J Gen Pract. 2015 Feb;65(631):101-2. doi: 10.3399/bjgp15X683665. No abstract available. PMID 25624305
- [Background] International working group of AAGL, ESGE, ESHRE and WES; Tomassetti C, Johnson NP, Petrozza J, Abrao MS, Einarsson JI, Horne AW, Lee TTM, Missmer S, Vermeulen N, Zondervan KT, Grimbizis G, De Wilde RL. An International Terminology for Endometriosis, 2021. J Minim Invasive Gynecol. 2021 Nov;28(11):1849-1859. doi: 10.1016/j.jmig.2021.08.032. Epub 2021 Oct 21. PMID 34690084
- See also: Menstrual Effluent Provides a Novel Diagnostic Window on the Pathogenesis of Endometriosis — https://doi.org/10.3389/frph.2020.00003
- See also: Single cell analysis of menstrual endometrial tissues defines phenotypes associated with endometriosis — https://doi.org/10.1101/2022.02.10.22270810
- See also: Analysis of menstrual effluent: diagnostic potential for endometriosis — https://doi.org/10.1186/s10020-018-0009-6

DOCUMENTS (1):
  • Study Protocol (2023-06-20): https://cdn.clinicaltrials.gov/large-docs/96/NCT05601596/Prot_000.pdf